CLINICAL TRIAL: NCT04178317
Title: Venetoclax (Venclexta Tablet) Post-Marketing Surveillance for CLL Patients
Brief Title: A Study of the Safety and Efficacy of Venetoclax for Participants With Chronic Lymphocytic Leukemia (CLL) Used in Routine Clinical Practice
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-942
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Cancer, Chronic Lymphocytic Leukemia (CLL)
Keywords: Cancer, Chronic Lymphocytic Leukemia (CLL), Venetoclax
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants receiving venetoclax for chronic lymphocytic leukemia according to the approved local label, and the decision to prescribe Venetoclax is independent from the enrollment into the study.

SUMMARY:
This observational study will evaluate the safety and effectiveness of Venetoclax used in routine clinical practice for participants diagnosed with chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with chronic lymphocytic leukemia who have been prescribed Venetoclax for the first time according to the approved label
* Participants (and/or legal representative) who voluntarily agree to participate in this study and sign informed consent

Exclusion Criteria:

-Participants with contraindications to venetoclax as listed on the approved local label

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Participants with chronic lymphocytic leukemia (CLL) who are prescribed venetoclax within the approved label according to physician judgement.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Up to Approximately 7 Years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either reasonable possibility or no reasonable possibility. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. For more details on adverse events please see the Adverse Event section.

SECONDARY OUTCOMES:
Overall Response | Up to Approximately 7 Years
  Overall Response will be assessed by the physician in charge of the study in accordance with the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- South Korea (13):
  - Inje University - Busan Paik Hospital /ID# 233882, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 216850, Busan, Busan Gwang Yeogsi
  - Kyungpook National University Hospital /ID# 233884, Daegu, Daegu Gwang Yeogsi
  - The catholic university of korea st. Paul's hospital /ID# 238907, Seoul, Gyeonggido
  - Ajou University Hospital /ID# 249512, Suwon, Gyeonggido
  - Chonnam National University Hwasun Hospital /ID# 216849, Hwasun-gun, Jeonranamdo
  - Korea University Anam Hospital /ID# 216851, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital /ID# 216853, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 217180, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 216852, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Seoul St. Marys Hospital /ID# 217181, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital /ID# 217179, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 215348, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info. — https://www.rxabbvie.com/